CLINICAL TRIAL: NCT03799757
Title: Role of Wound Installation With Bupivacaine Through Surgical Drains in Postoperative Analgesia in Modified Radical Mastectomy
Brief Title: Using Bupivacaine Locally in the Mastectomy Drains to Control Postoperative Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mahmoud A. Alhussini, lecturer surgical oncology, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: malhussini001
Record Dates: First submitted 2019-01-06; First posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Pain, Postoperative; Breast Cancer
Keywords: bupivacaine; Post-mastectomy acute pain; Wound instillation
MeSH Terms: conditions — Pain, Postoperative; Breast Neoplasms | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivacaine (Active Comparator): The wound was installed by 40ml of 0.25% bupivacaine through axillary and chest wall drains (20ml in each drain). Then, the drains were clamped for 20 minutes.
  Interventions: Drug: 40ml of 0.25% bupivacaine
- Placebo (Placebo Comparator): The wound was installed by 40ml of 0.9% normal saline through axillary and chest wall drains (20ml in each drain). Then, the drains were clamped for 20 minutes. (placebo group)
  Interventions: Drug: 40ml of 0.9% normal saline

INTERVENTIONS:
Drug: 40ml of 0.25% bupivacaine
  Arms: Bupivacaine
Drug: 40ml of 0.9% normal saline
  Arms: Placebo

SUMMARY:
in this study we are investigating the role of instillation of Bupivacaine through surgical drains at the end of mastectomy surgeries in controlling post operative pain and decreasing their pain killers requirement in the early postoperative period

DETAILED DESCRIPTION:
patients were enrolled into 2 groups. in one group the wound was installed by 40ml of 0.25% bupivacaine through axillary and chest wall drains (20ml in each drain). Then, the drains were clamped for 20 minutes.

in the other group the wound was installed by 40ml of 0.9% normal saline through axillary and chest wall drains (20ml in each drain). Then, the drains were clamped for 20 minutes. (placebo group) patients and health care providers were blinded as regard the study group patients enrolled in. Visual Analog Pain Scale which is a score for detection of how much the patient is annoyed from the pain- was assessed two and four hours post-operative then every four hours thereafter.

ELIGIBILITY:
Inclusion Criteria:

female patients with unilateral breast cancer candidates for total mastectomy and axillary dissection

Exclusion Criteria:

1. Male patients
2. Bilateral breast cancer.
3. Patients with a history of a long duration of NSAID intake or other painkillers, drug abuse
4. Patients with chest wall pain like Tietze syndrome, history of angina pectoris or recent HZV infection.
5. Patients with known psychological or mental problems.
6. Patients who were not exposed to axillary dissection

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only females with breast cancer who were subjected to mastectomy with axillary nodal dissection were enrolled
Enrollment: 168 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Visual analogue pain score | first 24 hours
  The intensity of pain will be assessed by the VAS score
Number of demands for analgesic | First 24 hours
  How many times the patient will require analgesics
Timing of first demand for analgesic | First 24 hours
  Time lapse between recovery from surgery and first demand for analgesic

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud A Alhussini, md, Principal Investigator — faculty of medicine , univeristy of alexandria
Locations (1):
- Faculty of Medicine, Main Univeristy Hospital, Alexandria, Egypt